CLINICAL TRIAL: NCT02671591
Title: A Pilot Study of PrEP Acceptance Among Young Black MSM
Acronym: MI-PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Crosby (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor-Investigator, Richard Crosby, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-02-10
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MI-PrEP (Experimental): This is a one-hour motivational interviewing-based, one-to-one session that will help YBMSM think more about going on PrEP. The control condition is a one-hour, theory-based, one-to-one session that will help YBMSM think more about using condoms consistently and correctly with every sex partner.
  Interventions: Behavioral: MI-PrEP
- control (Active Comparator): This condition will include the provision of free condoms and lubricants - selected from a buffet of condoms and lubricants designed to offer men a broad selection of high quality products that can optimize the "fit and feel" of condoms during sex.
  Interventions: Behavioral: control condition

INTERVENTIONS:
Behavioral: MI-PrEP — This is a one-hour motivational interviewing-based, one-to-one session that will help YBMSM think more about going on PrEP and it will help YBMSM think more about using condoms consistently and correctly with every sex partner.
  Arms: MI-PrEP
Behavioral: control condition — This is a behavioral program designed to provide men with condoms and lubricants that make sex feel good even though it is fully protected by latex condoms
  Arms: control

SUMMARY:
The overarching goal of the proposed study is to determine effective outreach methods designed to recruit and improve acceptance of high-risk HIV-negative YBMSM to initiate PrEP and to identify and modify psychosocial and structural predictors of PrEP acceptance. Specifically, the objective of this pilot study is to test the feasibility of a motivational interview-based intervention designed to improve PrEP acceptance among YBMSM.

DETAILED DESCRIPTION:
The study will occur in conjunction with standard clinical practice, which now includes offering high-risk YBMSM PrEP. If a person accepts this offer the person will be provided the service, but the person will not be asked to participate in the proposed study. Indeed, the study is designed for men who initially refuse this offer. Thus, for those who refuse researchers will offer study enrollment. For those who accept this offer and enroll, researchers will conduct baseline assessment and then randomize to I (intervention) versus C (control). Volunteers will receive the I or C condition immediately.

The intervention condition will be called MI-PrEP. This is a one-hour motivational interviewing-based, one-to-one session that will help YBMSM think more about going on PrEP. The control condition is a one-hour, theory-based, one-to-one session that will help YBMSM think more about using condoms consistently and correctly with every sex partner. This is the same program that is currently being tested at Crossroads, known as Focus on the Future. Both conditions (I and C) will include the provision of free condoms and lubricants - selected from a buffet of condoms and lubricants designed to offer men a broad selection of high quality products that can optimize the "fit and feel" of condoms during sex.

After receiving the I or C condition, researchers will collect extensive contact information for the volunteer and explain to the participant that researchers will make contact each week for the next 4 weeks, at which time researchers would like the participant to return to complete a second computer-assisted self-administered survey. Thus, approximately 4 weeks (but no later than six weeks) after study enrollment, the volunteer will return to the clinic for a second assessment. At this time, a second formal offer of PrEP by the clinician will be made (note: participants may accept the initial offer at any time up until this point). For persons accepting the offer of PrEP at this time, researchers will follow standard of care procedures and administer the PrEP. Nonetheless, this person will remain in study until 6 months has elapsed since enrollment occurred. At the conclusion of that 6-month period, blood will be collected to test for PrEP levels plus self-reported adherence measures will be collected and a follow-up computer-assisted self-interview will be given.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 29 years of age
* Identification as Black or African American
* Eligible for PrEP

Exclusion Criteria:

* none

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Decide to Take PrEP | 6 months
  Researchers will evaluate and compare the number of participants who decide to take PrEP in the control condition and MI-PrEP condition.

IPD SHARING:
Plan to Share IPD: No